CLINICAL TRIAL: NCT07287085
Title: Increasing Lung Cancer Screening Uptake Among Emergency Department Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Lung Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: FP 9214
Record Dates: First submitted 2025-12-02; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Screening Compliance; Lung Cancer (Diagnosis); Lung Cancer Diagnosis; Lung Cancer
Keywords: screening; lung cancer; screening compliance
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Basic Referral (enhanced control arm) (Active Comparator): Participants assigned to Arm 1 will be referred to the UR Medicine LCS Program and their primary care provider (if they have one) to discuss LCS. They will also be provided with written materials that include telephone contact information for the LCS Program Navigator.
  Interventions: Behavioral: Basic Referral (enhanced control arm)
- Facilitated Referral + Text Messaging (Experimental): For participants assigned to Arm 2, an LCS requisition form will be submitted to the UR Medicine LCS Program on behalf of the participant during their ED visit. The participant's primary care provider (if they have one) will be CC'd on the requisition. Participants will be instructed that the LCS program will reach out to them to discuss LCS and, if decided upon, schedule screening. An LCS Program Navigator will call the participant by phone, conduct a shared decision-making discussion, and schedule the screening CT scan (assuming eligibility is confirmed and the discussion results in the participant's decision to schedule screening). In addition, participants in Arm 2 will receive a series of text messages, grounded in the TPB, SDT, and HBM aimed at generating intention and motivation to get LCS.
  Interventions: Behavioral: Facilitated referral and text messaging

INTERVENTIONS:
Behavioral: Facilitated referral and text messaging — Participants randomized to the experimental arm will be instructed that the LCS program will reach out to them to discuss LCS and, if decided upon, schedule screening. An LCS Program Navigator will call the participant by phone, conduct a shared decision-making discussion, and schedule the screening CT scan (assuming eligibility is confirmed and the discussion results in the participant's decision to schedule screening). In addition, participants in Arm 2 will receive a series of text messages, grounded in the TPB, SDT, and HBM aimed at generating intention and motivation to get LCS.
  Arms: Facilitated Referral + Text Messaging
Behavioral: Basic Referral (enhanced control arm) — They will also be provided with written materials that include telephone contact information for the LCS Program Navigator. If contacted, the LCS Program Navigator will conduct a shared decision-making (SDM) discussion, schedule the screening CT scan at one of the 8 regional American College of Radiology-designated LCS centers and arrange follow-up as needed. Since determination of LCS needs is not routine during an ED visit, this "control arm" reflects an enhancement over usual care. It would not be ethical to identify a patient with screening needs without providing a referral.
  Arms: Basic Referral (enhanced control arm)

SUMMARY:
The objective of the proposed clinical trial is to determine if we can increase LCS among ED patients using a combination of facilitated referral to an LCS program plus text message reminders to get screened. Step 1 of the approach is to identify participants that are eligible for LCS. Step 2 is to randomize eligible study participants between two study arms: (1) basic referral for LCS (i.e.

verbal referral with written materials), and (2) facilitated referral for LCS (i.e. submission of a requisition to LCS program by staff) plus a subsequent series of text messages aimed at generating intention and motivation to get screened. The investigators' preliminary work showed this approach was feasible in the ED setting. The proposed study will build on this preliminary work with the goal of having a significant positive impact on LCS uptake.

A total of 300 individuals eligible for LCS will be recruited from a high-volume urban ED, randomized between study arms, and followed-up at 120 days to assess interval LCS uptake. The Specific Aims of the proposed project are, (1) Compare LCS uptake between the two study arms, (2) Identify predictors of individuals that are not up-to-date with LCS at the time of enrollment, and (3) Evaluate study participant feedback on (a) barriers and facilitators to getting screened and (b) acceptability and appropriateness of ED-based promotion of LCS. The study team is at the forefront of developing ED-based interventions to promote cancer screening. This project leverages the universal access setting of the ED to identify individuals at greatest risk for lung cancer and get them screened. A scalable ED-based intervention that increases LCS uptake would save lives.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 - 80
* ≥ 20 pack-year smoking history
* current smoker or quit within 15 years
* English speaking
* Current patient in URMC involved Emergency Department

Exclusion Criteria:

* Non-English
* Inability to provide consent (e.g. high clinical acuity, cognitive deficit)
* Lack of text-capable mobile phone and/or inability to use text function
* Not being a patient in URMC involved Emergency Department There are no restrictions for gender, racial and ethnic origins.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 349 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Assessment for LCS Uptake and Downstream Care | From enrollment through participation with first assessment at ~ 120 days of participation.
  The primary outcome, LCS uptake, will be assessed via telephone follow-up and EHR review.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided